CLINICAL TRIAL: NCT01228266
Title: Autologous Mesenchymal Stem Cell Transplantation in Multiple Sclerosis: a Randomized, Double-blind, Crossover With Placebo Phase II Study
Brief Title: Mesenchymal Stem Cell Transplantation in MS
Acronym: CMM-EM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Ended the recruitment in June 2012 for low enrollement accrual
Sponsor: Albert Saiz (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Albert Saiz, MD, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CMM-EM
Record Dates: First submitted 2010-10-25; First posted 2010-10-26 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- autologous mesenchymal stem cell (Experimental): A single infusion of up to 2 million cells per Kg of autologous mesenchymal stem cells vs suspension media. The treatment will be reversed at 6 months
  Interventions: Biological: autologous mesenchymal stem cells

INTERVENTIONS:
Biological: autologous mesenchymal stem cells — A randomized double-blind, crossover study comparing treatment with autologous MSC vs. suspension media on patients with active MS

SUMMARY:
The study is a randomized Phase II study, masked and crossed-over with placebo to evaluate the safety and tolerability of autologous mesenchymal stem cell transplantation in patients with active multiple sclerosis

ELIGIBILITY:
Inclusion Criteria:

1. Inflammatory forms of MS

   1. Relapsing-remitting MS (RRMS) patients
   2. Secondary progressive MS (SPMS) patients with continued relapses
   3. Primary progressive MS (PPMS) patients with enhancing MRI lesions and positive CSF (oligoclonal banding)
2. Age 18-50 years
3. Disease duration >= 2 and >= 10 years
4. EDSS 3.0 - 6.5
5. Progression, continued relapses or worsening MRI after at least a year of attempted therapy evidenced by:

   1. Increase of >= 1 EDSS point (if baseline EDSS <= 5.0) or 0.5 EDSS points (if baseline EDSS >= 5.5), or quantifiable, objective evidence of equivalent progression
   2. >= 1 moderate-severe relapses in past 18 months
   3. >= 1 Gadolinium enhancing lesions (double or triple dose Gadolinium)
   4. >= 1 new T2 lesion
   5. For PPMS only, >= 1 Gadolinium enhancing lesions
6. Has given informed consent to participate in the study.

Exclusion Criteria:

1. SPMS without ongoing relapses
2. PPMS without positive CSF or Gadolinium enhancing lesions
3. <= 3 months since treatment with any immunosuppressive therapy
4. <=1 month since last treatment with interferon-B or glatiramer acetate
5. Corticosteroid treatment <= 30 days
6. Relapse <= 60 days
7. History of cancer or clinical or laboratory results indicative of severe systemic diseases, including infection for HIV, Hepatitis B or C
8. Any metallic or electronic device that precludes from undergoing MRI
9. Pregnancy or lactation
10. Current treatment with an investigational therapy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2010-12; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety as number of severe events along 1 year, and efficacy in terms of cumulative number of gadolinium-enhancing lesions in MRI at 6 months and at the end of the study | 12 months
  The coprimary endpoints were safety and efficacy in terms of cumulative number of gadolinium-enhancing lesions in MRI

SECONDARY OUTCOMES:
To evaluate effects on MS disease activity measured by: clinical variables, MRI, OCT, immunological analysis and quality of life scales | 12 months
  clinical outcomes (number of relapses and change in the EDSS); MRI-based measures and OCT. Immunological evaluation as exploratory analysis

CONTACTS AND LOCATIONS:
Overall Officials: Albert Saiz, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Neurology Service, Hospital Clinic de barcelona, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Llufriu S, Sepulveda M, Blanco Y, Marin P, Moreno B, Berenguer J, Gabilondo I, Martinez-Heras E, Sola-Valls N, Arnaiz JA, Andreu EJ, Fernandez B, Bullich S, Sanchez-Dalmau B, Graus F, Villoslada P, Saiz A. Randomized placebo-controlled phase II trial of autologous mesenchymal stem cells in multiple sclerosis. PLoS One. 2014 Dec 1;9(12):e113936. doi: 10.1371/journal.pone.0113936. eCollection 2014. PMID 25436769